CLINICAL TRIAL: NCT06476925
Title: Role of Left Stellate Ganglion Block in Offering Myocardial Protection in On-pump Mitral Valve Replacement? A Histopathological and Clinical Assessment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1130/4/2024
Record Dates: First submitted 2024-06-18; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Open Mitral Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Sonar guided stellate ganglion injection of 8 ml of sterile saline 0.9% using high frequency probe as a placebo. Stellate ganglion is identified at the level of C6 just under the pulsation of the ipsilateral carotid artery
  Interventions: Procedure: sonar guided stellate ganglion injection
- Stellate ganglion (Active Comparator): Sonar guided stellate ganglion injection of 8ml bupivacaine 0.25% using high frequency probe. . Stellate ganglion is identified at the level of C6 just under the pulsation of the ipsilateral carotid artery
  Interventions: Procedure: sonar guided stellate ganglion block

INTERVENTIONS:
Procedure: sonar guided stellate ganglion injection — using high frequency probe, sonar guided stellate ganglion block with 8 ml saline 0.9%
  Arms: Control group
Procedure: sonar guided stellate ganglion block — using high frequency probe, sonar guided stellate ganglion block with 8 ml bupivacaine 0.25%
  Arms: Stellate ganglion

SUMMARY:
Can pre-operative left stellate ganglion block offer myocardial protection in on-pump mitral valve replacement? A histopathological and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult population of both sex, between 25-50 years, will undergo elective on pump mitral valve replacement

Exclusion Criteria:

* -Combined valve replacement ( mitral and aortic or mitral and tricuspid valves replacement).
* Emergency valve replacement ( stuck valve, infective endocarditis).
* Pre-operative cardiomyopathy (Ejection fraction less than 45%).
* Recent myocardial infarction ( within 6 months)
* Redo mitral valve replacement.
* Pre-operative pacing, or cardioverter, any form arrhythmia ( tachy or brady).
* Previous history of carotid endarterectomy or presence of carotid stent.
* On thrombolytic therapy.
* Severe chronic obstructive airway disease,
* Patient refusal

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with microscopic myocardial injury | intra-operative
  Biopsy from left papillary muscle to investigate microscopic evidence of cellular injury ( cytoplasmic oedema, hemorrhage and necrosis).

SECONDARY OUTCOMES:
Intra-operative arrhythmia | intraoperatively
  incidence of intraoperative atrial fibrillation
postoperative arrhythmia | first, second and third day after bypass
  Incidence of post operative atrial or ventricular arrhythmia
Troponin I | before operation, immediately after ICU admission and 3 days post-operative
  Serum troponin I to diagnose myocardial injury
Myocardial function | pre-operative, one week
  Ejection fraction
weaning from mechanical ventilation | 24 hours post-operative
  Time from ICU admission till successful extubation
Time of cardiopulmonary bypass | Intraoperative
Length of ICU stay | one week
Need for pacing | intraoperative and one week after